CLINICAL TRIAL: NCT00398424
Title: A Phase I, Open-Label Study Evaluating The Pharmacokinetics of Components of S-1 Patients With Impaired Hepatic Function
Brief Title: Evaluating Patients With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Peter Urrea/Senior VP Clinical and Regulatory Affairs, Taiho Pharma USA, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1112
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Impaired Hepatic Function
Keywords: Impaired Hepatic Function
MeSH Terms: interventions — S-1 plus cisplatin

INTERVENTIONS:
Drug: S-1/Cisplatin — PK Phase (Part 1), Beginning on Day 1 of the Pharmacokinetic Phase, 30 mg/m2 S-1 will be administered orally BID for 14 days (Days 1 through 14), followed by a 1-week recovery period.
  On Day -2 and Day 14 of the Pharmacokinetic Phase, all patients will receive a single dose of 30 mg/m2 S-1 administered orally.
  Extension Phase, Patients will receive S-1 at the dose that they tolerated in the PK Phase. S-1 will be administered orally BID for 2 weeks (Day 1 through Day 14) followed by a 1-week recovery period (Day 15 through Day 21). This cycle will be repeated every 3 weeks.

SUMMARY:
This is a Phase I, Open-Label study evaluating the PK of S-1 components and their metabolites in patients with advanced solid tumors and varying degrees of hepatic function defined by the NCI classification for hepatic impairment. Patients will be stratified into 4 Cohorts- Normal, Mild, Moderate or Severe.

Six patients will be enrolled inot each cohort and receive S-1.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. Has histologically or cytologically proven advanced solid tumors for which no standard therapy exists.
2. Has provided written informed consent.
3. Is 18 years of age or older.
4. Is able to take medications orally.
5. Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to ≤ 2 (Appendix A, ECOG Performance Status).
6. Has adequate organ function as defined by the following criteria:

   1. Absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units [IU]).
   2. Has a platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
   3. Has a hemoglobin value of ≥ 9.0 g/dL.
   4. Has a calculated creatinine clearance > 60 mL/min (by Cockcroft-Gault
7. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria

Exclude a patient from this study if he/she does not fulfill the inclusion criteria, or if any of the following conditions are observed:

1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Any investigational agent received either concurrently or within the last 30 days.
   2. Previous therapy for malignancy within 21 days, including any chemotherapy, immunotherapy, biologic or hormonal therapy (6 weeks for nitrosoureas or mitomycin C).
   3. Previous radiotherapy within 14 days.
   4. Current enrollment in another clinical trial.
   5. Required shunting or stenting of the liver within prior 28 days or planned during the first study treatment cycle.
2. Has a serious illness or medical condition(s) including, but not limited to, the following:

   1. Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure (New York Heart Association [NYHA] Class III or IV, see Appendix F, NYHA Classification).
   2. Known (at the time of entry) gastrointestinal disorder, including malabsorption,chronic nausea, vomiting, or diarrhea present to the extent that it might interfere with oral intake and absorption of the study medication.
   3. Previous organ allograft, including liver transplantation.
   4. Known brain metastasis.
   5. Known leptomeningeal metastases.
   6. Manifest ascites.
   7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
   8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study. • 3. Is receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

   <!-- -->

   1. Sorivudine, uracil, dipyridamole, cimetidine and folinic acid (may enhance S-1 activity).
   2. Allopurinol (may diminish S-1 activity).
   3. Phenytoin (S-1 may enhance phenytoin activity).
   4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 and flucytosine activity).
   5. Pilocarpine (may inhibit CYP2A6 activity).

4. Has known sensitivity to 5-FU. 5. Is a pregnant or lactating female. 6. Is a patient with reproductive potential who refuses to use an adequate means of contraception (including male patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To provide specific dosing recommendations for S-1 in patients with hepatic impairment based on the PK of S-1 and its components after single dose and during steady state condition | The Pharmacokinetic Phase (Part 1) of the study will last 24 days.

SECONDARY OUTCOMES:
To assess the antitumor activity and safety profile of S-1 in patients with impaired hepatic function | Each cycle of the Extension Phase (Part 2) will be 21 days (14 days of S-1 treatment, 7 days recovery). The end of study for the Extension Phase will be 30 days after the last dose of S-1.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - University of Kentucky/Division of Hematology/Oncology and Blood Marrow Transplantation, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - The Institute for Drug Development, San Antonio, Texas